CLINICAL TRIAL: NCT02363036
Title: The Shift From Monocytes to Neutrophils in Blood Samples of Women in Labor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0004-15-HYMC
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-01

CONDITIONS: Parturition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Active labor: Women in active labor normal pregnancy at term.
- Planned Cesarian Section: Women, normal pregnancy at term who came for elective Cesarean Section without signs of labor (pain/contractions, etc).

SUMMARY:
Accumulating evidence suggest that the proliferative, invasive, and immune tolerance mechanisms that malignant tumors use to establish a nutrient supply and evade or edit the host immune response are similar to those used by the developing placenta during normal pregnancy. In addition to the shared capacity for invading through normal tissues, both cancer cells and cells of the developing placenta create a microenvironment supportive of both immunologic privilege and angiogenesis.

CD11b+Gr1+ cells are a heterogeneous population of bone marrow-derived cells (BMDC) that consist of immature myeloid cells (IMCs), and were first described as myeloid-derived suppressor cells. In healthy individuals, IMCs that are generated in the bone marrow differentiate into mature granulocytes, macrophages, or dendritic cells (DCs). These cells have been shown to play an essential role in mediating immune suppression in animal models of human tumors. As a result of tumor-induced alterations in myelopoiesis, IMCs have been found in peripheral blood, lymphoid organs and the tumor tissue itself. An increased population of IMCs was identified in patients with several tumor types. Accordingly, IMCs detected in the peripheral blood of such patients bearing express the common myeloid marker CD33 but lack markers of mature myeloid cells such as the MHC class II molecule HLADR.

IMCs have been shown to actively promote tumor growth and metastasis by modulating the cytokine environment, and through vascular remodeling by promoting angiogenesis.

It has been demonstrated in our laboratory that IMCs infiltrate placentas of pregnant mice and actively promote angiogenesis. These cells show striking similarity to IMCs that populate malignant tumors. Accordingly, human placentas are also infiltrated by a significant population of IMCs. Immunostaining of human placentas showed that IMCs comprise around 25% ( range 10-40%) of total placental CD45+ bone marrow-derived hematopoietic cells and that this population is located close to blood capillaries. We also demonstrated that immature DCs, cells originally described to regulate the adaptive immune response, also promote angiogenesis in models of choroidal neovascularization, endometriosis and tumors.

This is a retrospective study on patient's blood samples of pregnant women who came to delivery in our department during 1.1.2014-31.12.2014, to compare the abundance of monocytes and neutrophils in: 1. Term active labor. 2. Elective cesarean section.

According to our previous findings, we hypothesize that monocytes in active delivery will be lower than in women without signs for labor. We also hypothesize that neutrophils will be more abundant in active delivery than in women without signs for labor.

We plan to screen anonymous electronic data of women who delivered in our departement during 2014 according to the following eligible criteria, stratified into 2 categories: 1. Women who were admitted in active labor. 2. Women who were admitted for elective Cesarean Section without signs of labor.

We will compare the abundance of monocytes and neutrophils in blood counts that were taken on admission day between the two populations.

ELIGIBILITY:
Inclusion Criteria:

* Women in active labor normal pregnancy at term.
* Women, normal pregnancy at term who came for elective Cesarean Section without signs of labor (pain/contractions, etc).

Exclusion Criteria:

* Signs for infection ( fever >38 celsius degrees)
* Women in pre-term birth under 37 weeks.
* Any complication to the women or fetus which require induction of labor ( Pre-eclampsia, Gestational Diabetes Mellitus A2, Pre-gestational diabetes, Intrauterine Growth Restriction).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy women without any complications in the current pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Delivery | 24 hours
  From admission time to delivery